CLINICAL TRIAL: NCT04827797
Title: Effects of Different Birthing Balls Used at the First Stage of Childbirth on Birth Outcomes and Maternal Satisfaction November, 2018
Brief Title: Effects of Different Birthing Balls Used at the First Stage of Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Tugce Sonmez, Principal Investigator, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 3301cukurova
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Labor Pain; Satisfaction, Patient; Labor Fast
Keywords: birth ball; labor pain; satisfaction; maternal; fetal
MeSH Terms: conditions — Labor Pain; Patient Satisfaction; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- birth ball (Experimental): The positions and movements for birth ball in the active and latent phases: kneeling on the ground and leaning on the spherical birthing ball, sitting on the ball with front support, sitting positions on the spherical birthing ball, full rotation of hip, moving to the right/left, back and forth. Positions and movements were repeated every 30 minutes. The 30-minute intervals were interrupted in cases where the women were not feeling well.
  Interventions: Device: balls
- peanut ball (Experimental): The positions and movements for the pregnant women in peanut ball: upright sitting position, forward bending positions, with backward and forward movement and swaying right and left on the peanut ball
  Interventions: Device: balls

INTERVENTIONS:
Device: balls — Birth balls to exercise
  Other Names: Birth ball; Peanut Ball

SUMMARY:
The study aimed to determine the effects of different birthing balls used at the first stage of childbirth on birth outcomes and maternal satisfaction. Randomized controlled, single-blind clinical study included a total of 180 pregnant women. The study included 3 groups (A: routine hospital care, B: spherical birthing ball, C: peanut ball). Especially spherical birthing ball, were effective in reducing labor pain and facilitating faster rate of descent of the fetal head, and they increased maternal satisfaction.

DETAILED DESCRIPTION:
The study aimed to determine the effects of different birthing balls used at the first stage of childbirth on birth outcomes and maternal satisfaction. Randomized controlled, single-blind clinical study included a total of 180 pregnant women. The study included 3 groups (A: routine hospital care, B: spherical birthing ball, C: peanut ball). Especially spherical birthing ball, were effective in reducing labor pain and facilitating faster rate of descent of the fetal head, and they increased maternal satisfaction.

IMPACT STATEMENT What is already known on this subject? Labor pain and outcomes occurring during labor are known and expected situation. Some non-pharmacological methods are applied to ensure that birth is easy and maternal satisfaction is high.

What the results of this study add? There is no studies using the peanut ball and the spherical birth ball together. In our study, it was found that both balls are effective, but the spherical birth ball is more significant.

What the implications are of these findings for clinical practice and/or further research? Our study suggested that the spherical birth ball had effective on birth outcomes. Future studies should be performed to investigate the effects of birth balls in the postpartum period, breastfeeding or prenatal period.

ELIGIBILITY:
Inclusion Criteria:

* primiparous
* admitted to the delivery room for vaginal delivery
* 38-40 week
* being in the latent phase of labor
* having no obstetric risks

Exclusion Criteria:

* undergo caesarean sections for various reasons
* having obstetric risks

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | when pregnant women come to the delivery room
  this form consists of 7 questions regarding participants' descriptive and obstetric characteristics.
Visual Analogue Scale | Latent, active and transition phase in labor
  in this scale, the participants marked the severity of their pain on a 10-cm ruler with one end stating "no pain" and the other end "worst possible pain". VAS was used to determine the severity of pain and the effectiveness of the intervention in this study.
Verbal Rating Scale | Latent, active and transition phase of labor
  This scale is based on participants' choice of word that defines their pain state
Partogram | active phase of labor
  This is used starting from the active phase of labor. The progress of the labor and the health status of the baby are monitored on the partogram
Evaluation Scale for Maternal Satisfaction with Normal Delivery | within a period of 1-4 hours postpartum
  This is used to assess maternal satisfaction in normal delivery. Higher total scores on the scale indicate stronger maternal satisfaction with the hospital care provided in normal delivery

CONTACTS AND LOCATIONS:
Overall Officials: tuğçe sönmez, Principal Investigator — Gaziantep ıslamic science and tecnology university
Locations (1):
- Tuğçe Sönmez, Toroslar, Mersin, Turkey (Türkiye)